CLINICAL TRIAL: NCT03072784
Title: Implication of Aortic Cross Clamping Time Upon Postoperative Respiratory Function in Adult Patients Undergoing Open Heart Surgery
Brief Title: Aortic Cross Clamping Time, and Postoperative Respiratory Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Lecturer of Anesthesia and critical care Medicine, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB00009915
Record Dates: First submitted 2017-02-15; First posted 2017-03-07 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Bypass Complication; Respiratory Complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group S (Active Comparator): short time <90 m aortic cross clamping
  Interventions: Procedure: aortic cross clamping
- group L (Active Comparator): > 90 minutes aortic cross clamping
  Interventions: Procedure: aortic cross clamping

INTERVENTIONS:
Procedure: aortic cross clamping — duration of cross clamping, less than 90 minutes, or more than 90 minutes

SUMMARY:
Does the duration of cardiopulmonary bypass, and aortic cross clamping affects the post operative pulmonary function.

DETAILED DESCRIPTION:
Cardiac surgery usually is done under cardiopulmonary bypass. As the blood contacts with the artificial tubing of the circuit, there is release of mediators which affects pulmonary function. Of no doubt that the duration of cardiopulmonary bypass, and cross clamping time, will affect the spell over of such mediators. Follow up of the pulmonary function, and arterial blood gas is mandatory in such group of patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* elective open heart surgery

Exclusion Criteria:

* Patients with myocardial ischemia or previous infarction
* low ejection fraction <30%
* history of AF
* implanted pacemaker
* uncontrolled hypertension
* renal impairment (creatinine >1.8 mg/dl)
* hepatic dysfunction
* insulin dependent diabetes
* chronic pulmonary disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-04-20 (Actual); Study Completion 2016-08-25 (Actual)

PRIMARY OUTCOMES:
quality of oxygenation | 48 hours postoperative
  PaO2 mmHg

SECONDARY OUTCOMES:
time to extubation | 24 hours postoperative
  time to extubate in minutes
ventilation | 48 hours postoperative
  respiratory rate (breath/minute)
carbon dioxide | 48 hours
  PaCO2 mmhg

CONTACTS AND LOCATIONS:
Overall Officials: Emad Z kamel Said, MD, Principal Investigator — Assiut University
Locations (1):
- Emad Zarief Kamel Said, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided